CLINICAL TRIAL: NCT02117323
Title: Observational Study on Corneal Opacities in Children
Brief Title: Corneal Opacities in Children
Acronym: OCT
Status: Completed | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, David Huang, David Huang, MD, PhD, Weeks Professor of Ophthalmology, Oregon Health and Science University, Oregon Health and Science University
Other Study IDs: CCI-10-00084; R01EY018184 (NIH)
Record Dates: First submitted 2014-01-14; First posted 2014-04-17 (Estimated); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Corneal Opacities
Keywords: corneal opacities; Optical coherence tomography
MeSH Terms: conditions — Corneal Opacity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
A prospective observational study on corneal opacities in infants and children (1 month to 18 years old) will be conducted at CHLA. Most of these cases will be due to congenital corneal opacity (e.g. Peter's anomaly, mucopolysacharidoses) or scarring due to infectious keratitis. Sixty (60) subjects will be recruited. The children will be examined under anesthesia with a portable slit-lamp and OCT. An iVue OCT system (Optovue) attached to an operating microscope-style mount at CHLA will be used for the intraoperative scans. Both cross-sectional and 3-D OCT scans will be performed to assess opacity depth, pachymetry map, endothelial defects, and any abnormal adhesion between the cornea, iris and lens. The anterior chamber angle will also be imaged with cross-sectional OCT to assess angle depth, trabecular meshwork, Schwalbe's line, and possible peripheral iridocorneal adhesion or posterior embryotoxon. OCT of the crystalline lens will be obtained to assess the presence of cataract. Slit-lamp photography will be obtained, and gonioscopy will be performed if indicated. Corneal diameter will be measured with a caliper, and intraocular pressure will be measured with a tonopen (Reichert).

ELIGIBILITY:
Inclusion Criteria:

* Infants and children (1 month to 18 years of age) with corneal opacity requiring a thorough eye examination.

Exclusion Criteria:

* Inability to give informed consent.
* Inability to maintain stable fixation for OCT imaging.
* Inability to commit to required visits to complete the study.

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Infants and children (1 month to 18 years of age) with corneal opacity requiring a thorough eye examination.
Sampling Method: Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2011-09; Primary Completion 2016-08-31 (Actual); Study Completion 2016-08-31 (Actual)

PRIMARY OUTCOMES:
Number of suitable subjects | 5 years
  The primary goal of the study will be to identify subjects suitable for the trial with OCT-guided LALAK. The determination will be based on analysis of clinical history & OCT corneal images as well as the subjects' willingness to participate in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Bibiana Reiser, MD, Principal Investigator — Children's Hospital Los Angeles
Locations (1):
- Children's Hospital Los Angeles, Los Angeles, California, United States